CLINICAL TRIAL: NCT02579642
Title: Effects of Low-dose Ketamine as an Adjunct to Propofol-based Anesthesia for Electroconvulsive Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Ferrante Gragasin, Associate Clinical Professor and Postgraduate Research Director, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00044771
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Depressive Disorder
Keywords: Moderate to severe depression; Monopolar; Bipolar; Ketamine; ECT; Electroconvulsive therapy; NMDA
MeSH Terms: conditions — Depressive Disorder | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Propofol at usual induction doses for ECT (0.75 - 1 mg/kg IV bolus) with placebo (normal saline)
  Interventions: Drug: Placebo
- Ketamine (Experimental): Propofol at usual induction doses for ECT (0.75 - 1 mg/kg IV bolus) with the addition of low-dose ketamine 0.2 mg/kg (or 0.5 mg/kg - see interim analysis)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Low dose ketamine 0.2 mg/kg (or 0.5 mg/kg depending on results of interim analysis) administered with usual induction drugs for ECT
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Normal saline administered with usual induction drugs for ECT
  Other Names: Normal saline; 0.9% NS
  Arms: Placebo

SUMMARY:
Ketamine has been used successfully as the sole medication for anesthesia in the setting of electroconvulsive therapy (ECT), and has more recently been studied as an adjunct agent in combination with propofol (the most commonly used anesthetic agent) to induce anesthesia for ECT. New literature postulates an anti-depressant effect of ketamine, which in ECT specifically may be helpful with regards to the overall goals of therapy (i.e. ECT indicated for severe or treatment-resistant depression).

Current research focusing on ketamine with respect to its anti-depressant effect suggests it may even represent an alternative to ECT. This study will seek to determine whether ketamine when used in low-doses as an adjunct to propofol-based anesthesia for ECT has anti-depressant effects and whether it influences the characteristics of recovery from anesthesia in the ECT setting (i.e. vital sign parameters such as blood pressure and heart rate, quality of recovery, etc.).

DETAILED DESCRIPTION:
This is a proof-of-concept study to elucidate whether the use of low-dose ketamine as an adjunct to propofol-based anesthesia for electroconvulsive therapy has beneficial anti-depressant effects in a population of adults with major depressive disorder presenting for ECT.

Since thiopental is no longer widely available in North America as an induction agent for anesthesia, other agents have supplanted it for various uses, including for induction of anesthesia for electroconvulsive therapy (ECT). Induction is most commonly achieved using propofol in doses of 0.75 - 1 mg/kg IV bolus.

Propofol as an induction agent for ECT may not be the ideal agent in this setting as its anticonvulsant effects may result in less-than-ideal seizure quality and duration. Ketamine has been studied in the ECT setting but at full induction doses has well-known psychotomimetic and dissociative effects. However, the anti-depressant effects of ketamine, even at low-doses, may have a beneficial effect on depressive symptoms after ECT as compared with propofol alone.

Ketamine also has been used successfully as the sole induction agent for anesthesia in this setting, and has more recently been studied as an adjunct or co-induction agent in combination with propofol. Drawbacks of using ketamine as the sole induction agent are related to its hemodynamic and psychotomimetic effects (e.g. post-treatment hypertension and hallucinogenic activity).

New literature postulates a putative anti-depressant effect of ketamine via the N-Methyl-D-aspartate (NMDA) receptor, which in the ECT setting specifically may be helpful with regards to the overall goals of therapy (i.e. ECT indicated for severe or treatment-resistant depression). Current research focusing on the efficacy of ketamine with respect to anti-depressant effects suggests that ketamine may even represent an alternative to ECT.

As per the investigators' standard practice for ECT, treatment for each patient would be 3 times per week up to a total of 12 treatments (i.e. 4 weeks of treatment). The total study duration for each patient will be not more than 6 weeks. As discussed below, patients will be withdrawn from the study at anytime upon their own request or when the treating psychiatrist feels the clinical improvement is strong enough to justify doing so.

An interim analysis will be completed after the first 14 patients have completed treatment. If after these first 14 patients the investigators find a lower than expected difference in efficacy in favor of the ketamine group, able to achieve alpha error >0.2 and power <80%, all subsequently recruited patients will be randomized to receive either propofol at usual induction doses for ECT (0.75 - 1 mg/kg IV bolus) with placebo (normal saline), or with a slightly higher dose of ketamine of 0.5 mg/kg. Should this turn out to be the case, thirty new patients will be recruited from that point.

ELIGIBILITY:
Inclusion Criteria:

* referred for ECT with a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of major depressive disorder
* considered American Society of Anesthesiologists (ASA) Physical Class I - III
* baseline MADRS score greater than 24 (i.e. at least moderate to severe depression)
* a "first" or "new" episode of depression which has lasted not more than 3 months and requires ECT treatment as judged by a psychiatrist

Exclusion Criteria:

* ASA Class IV or V as judged by the anesthesiologist
* Any ECT treatment in the previous three months
* Inability or refusal to provide informed consent
* A history of allergic reactions, hypersensitivity, or intolerance to anesthetics or their constituents used in the study (ketamine, propofol, egg phosphatide, soybean oil)
* Anyone taking medications considered contraindicated for ECT or for general anesthesia
* Presence of any of the following DSM-IV diagnoses: Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), abuse of opiates, amphetamines, barbiturates, cocaine, cannabis, or hallucinogen abuse in the 4 weeks prior to enrolment, pervasive developmental disorder, dementia
* Significant medical condition that would contraindicate the use of ketamine, propofol or that is untreated and would need urgent attention (as determined by treating physician)
* Medical conditions that would significantly affect absorption, distribution, metabolism, or excretion of ketamine or propofol
* Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
* Patients with increased risk of laryngospasm (such as active pulmonary infection, upper respiratory infection, asthma), increased intracranial pressure, glaucoma, thyroid disease/hyperthyroidism
* Any clinically significant deviation from the reference range in clinical laboratory test results as judged by the investigator
* Pregnancy (or female of child-bearing age not using adequate contraception) or lactation
* Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Number of treatments to achieve 50% change (reduction) in Montgomery Ashberg Depression Rating Scale (MADRS) | 6 weeks
  Defined a priori as "response". Assessed at baseline, 24 hours after ECT treatments for the duration of the study and then once at 6 weeks.

SECONDARY OUTCOMES:
Number of treatments to achieve 25% change (reduction) in MADRS | 6 weeks
  Defined a priori as "partial response". Assessed at baseline, 24 hours after ECT treatments for the duration of the study and then once at 6 weeks.
Change in Clinical Global Impression - Severity (CGI-S) scores | 6 weeks
  Assessed at baseline, 24 hours after ECT treatments for the duration of the study and then once at 6 weeks.
Changes in blood pressure seen during ECT | 4 weeks
  Measured during ECT treatments and in the post-ECT recovery room.
Changes in heart rate seen during ECT | 4 weeks
  Measured during ECT treatments and in the post-ECT recovery room.
Changes in oxygen saturation seen during ECT | 4 weeks
  Measured during ECT treatments and in the post-ECT recovery room.
Changes in respiratory rate seen during ECT | 4 weeks
  Measured during ECT treatments and in the post-ECT recovery room.
Changes in times to discharge from post-ECT recovery | 4 weeks

OTHER OUTCOMES:
Changes in seizure duration during ECT | 4 weeks
  As measured by clinical/visual assessment as well as by EEG.

CONTACTS AND LOCATIONS:
Overall Officials: Ferrante S Gragasin, MD, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Hospital Edmonton, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

REFERENCES:
- [Background] Okamoto N, Nakai T, Sakamoto K, Nagafusa Y, Higuchi T, Nishikawa T. Rapid antidepressant effect of ketamine anesthesia during electroconvulsive therapy of treatment-resistant depression: comparing ketamine and propofol anesthesia. J ECT. 2010 Sep;26(3):223-7. doi: 10.1097/YCT.0b013e3181c3b0aa. PMID 19935085
- [Background] Wang X, Chen Y, Zhou X, Liu F, Zhang T, Zhang C. Effects of propofol and ketamine as combined anesthesia for electroconvulsive therapy in patients with depressive disorder. J ECT. 2012 Jun;28(2):128-32. doi: 10.1097/YCT.0b013e31824d1d02. PMID 22622291
- [Background] Larkin GL, Beautrais AL. A preliminary naturalistic study of low-dose ketamine for depression and suicide ideation in the emergency department. Int J Neuropsychopharmacol. 2011 Sep;14(8):1127-31. doi: 10.1017/S1461145711000629. Epub 2011 May 5. PMID 21557878 (Retraction: PMID 28637184 Int J Neuropsychopharmacol. 2017 Jul 1;20(7):611)
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Derived] Woolsey AJ, Nanji JA, Moreau C, Sivapalan S, Bourque SL, Ceccherini-Nelli A, Gragasin FS. Low-dose ketamine does not improve the speed of recovery from depression in electroconvulsive therapy: a randomized controlled trial. Braz J Psychiatry. 2022 Jan-Feb;44(1):6-14. doi: 10.1590/1516-4446-2020-1705. PMID 34076068